CLINICAL TRIAL: NCT06586294
Title: A Phase Ib/II Open Label,Dose Escalation and Dose Extension Study Evaluating the Safety, Tolerability, and Initial Antitumor Efficacy of Anti-PD-1 and Lymphocyte Activation Gene 3(LAG-3) Bispecific Antibody AK129 Combined With Chemotherapy With or Without Cadonilimab in Patients With Human Epidermal Growth Factor Receptor 2 (HER2) Negative Unresectable Locally Advanced or Metastatic G/GEJ Adenocarcinoma
Brief Title: A Study of Anti-PD-1 and LAG-3 Bispecific Antibody(AK129) Combined With Chemotherapy With or Without Cadonilimab in the First-line Treatment of Unresectable Locally Advanced or Metastatic G/ GEJ Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK129-103
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Phase 1b/II, open-label, 2-part, multicenter, non-randomized, multiple-dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The dose escalation and expansion stage of AK129 combined with chemotherapy; (Experimental): Part 1: The dose escalation stage： 3 dose groups of AK129 were set up, combination with chemotherapy of XELOX,followed by AK129 and capecitabine maintenance; Part 2：The dose expansion stage： Two to three dosing regimens were set for expansion of AK129 in combination with XELOX.
  Interventions: Drug: Drug: AK129 Drug：oxaliplatin Drug：capecitabine
- The dose escalation and expansion stage of AK129 combined with chemotherapy with cadonilimab (Experimental): Part 1:The dose escalation stage： 3 dose groups of AK129 were set up, combination with cadonilimab and chemotherapy of XELOX,followed by AK129 and cadonilimab maintenance; Part 2:The dose expansion stage： Two to three dosing regimens were set for expansion of AK129 in combination with cadonilimab and chemotherapy of XELOX.
  Interventions: Drug: Drug: AK129 Drug：cadonilimab Drug：oxaliplatin Drug：capecitabine

INTERVENTIONS:
Drug: Drug: AK129 Drug：oxaliplatin Drug：capecitabine — AK129 is administered intravenously according to the frequency every three weeks(Q3W) and different dosage of administration at different stages.Oxaliplatin is administered intravenously according to the frequency and dosage 130 mg/m2 on day 1 Q3W.Capecitabine is administered intravenously according to the frequency and dosage 1000 mg/m2 oral twice daily on day 1 to 14 Q3W.
  Arms: The dose escalation and expansion stage of AK129 combined with chemotherapy;
Drug: Drug: AK129 Drug：cadonilimab Drug：oxaliplatin Drug：capecitabine — AK129 is administered intravenously according to the frequency Q3W and different dosage of administration at different stages. Cadonilimab is administered intravenously according to the frequency and dosage 10mg/kg Q3W.Oxaliplatin is administered intravenously according to the frequency and dosage 130 mg/m2 on day 1 Q3W.Capecitabine is administered intravenously according to the frequency and dosage 1000 mg/m2 oral twice daily on day 1 to 14 Q3W.
  Arms: The dose escalation and expansion stage of AK129 combined with chemotherapy with cadonilimab

SUMMARY:
Phase Ib/II clinical study of AK129 combined with chemotherapy with or without cadonilimab in first-line treatment of advanced HER2 negative gastric cancer or gastroesophageal junction adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the written informed consent form(ICF) voluntarily.
2. Aged ≥ 18 to ≤ 75 years,male and female at the time of signing the ICF.
3. Histologically confirmed adenocarcinoma of the gastric or gastroesophageal junction (GEJ).
4. Inoperable locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma.
5. Participants had not previously received systemic therapy for locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma.
6. According to RECIST v1.1 criteria, subjects had at least one measurable tumor target.

Exclusion Criteria:

1. Subjects with known HER2 positive gastric or gastroesophageal junction adenocarcinoma.
2. Histopathological examination confirmed other pathological types.
3. Had received palliative local therapy for non-target lesions within 2 weeks before the first administration.
4. Past treatment with immune checkpoint inhibitors,immune checkpoint agonists,immune cell therapy and any treatment targeting the immune mechanism of tumor action.
5. History of gastrointestinal perforation and fistula within 6 months before the first dose.
6. Active or previously documented inflammatory bowel disease,inability to swallow, malabsorption syndrome.
7. Active malignancy within the last 3 years.
8. Active or untreated brain metastases, meningeal metastases, spinal cord compression, or pia meningeal disease are known to exist.
9. The presence of clinical symptoms of pleural effusion, pericardial effusion, or abdominal effusion, or the need for frequent drainage.
10. There was an active autoimmune disease that required systemic treatment within 2 years prior to the start of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events(AE) | Up to approximately 2 years
  Incidence and severity of AEs is aim to evaluate the safety of AK129 combined with chemotherapy with or without cadonilimab
Incidence of serious adverse events(SAE) and suspected unexpected serious adverse reactions(SUSAR) | Up to approximately 2 years
  Incidence of SAE and SUSAR is aim to evaluate the safety of AK129 combined with chemotherapy with or without cadonilimab
Incidence of dose-limiting toxicity(DLT) | Up to approximately 2 years
  The purpose of DLT is to find the Phase II recommended dose(RP2D) or Maximum Tolerated Dose(MTD)
Clinically significant changes in safety/laboratory evaluation parameters and AEs that led to treatment termination or suspension | Up to approximately 2 years
  Clinically significant changes in safety/laboratory evaluation parameters and AEs that led to treatment termination or suspension is aim to evaluate the safety of AK129 combined with chemotherapy with or without cadonilimab
Objective Solution Rate (ORR) based on RECIST v1.1 | Up to approximately 2 years
  The purpose of ORR is aim to evaluate the antitumor effect,and ORR is proportion of subjects with complete response(CR) or partial response(PR), based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1.

SECONDARY OUTCOMES:
Disease control rate(DCR) | Up to approximately 2 years
  Disease control rate(DCR) is defined as the proportion of subjects achieving a best of response(BOR) of confirmed CR or PR or stable disease(SD) per RECIST v1.1.
duration of response(DoR) | Up to approximately 2 years
  Duration of response(DoR) is defined as the period from the first documentation of confirmed response(CR or PR) to the first documentation of progressive disease(PD) as per RECIST v1.1 or death due to any cause, whichever occurs first.
time to response(TTR) | Up to approximately 2 years
  Time to response(TTR) is defined as the time from the first dose of investigational products until the first confirmation of CR or PR.
progression-free survival(PFS) | Up to approximately 2 years
  Progression-free survival(PFS) is defined as the time from the first dose of investigational products until documentation of progressive disease(PD) as per RECIST v1.1 or death due to any cause, whichever occurs first.
overall survival(OS) | Up to approximately 2 years
  Overall survival(OS) is defined as the time from the first dose of investigational products until death due to any cause.
Serum AK129, cadonilimab concentration, blood concentration-time curve and derived PK argument | Up to approximately 2 years
  Serum AK129, cadonilimab concentration, blood concentration-time curve and derived PK argument to evaluate the Pharmacokinetics(PK).
Number and percentage of subjects with anti-drug antibodies (ADA) for AK129 and cadonilimab | Up to approximately 2 years
  Number and percentage of subjects with anti-drug antibodies (ADA) for AK129 and cadonilimab will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No